CLINICAL TRIAL: NCT03170973
Title: Influences of Physical Activity in the Profile of Trans Fatty Acids in the Serum of Individuals With Body Weight Changes
Brief Title: Influence of Exercise on Trans Fatty Acids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculdade Adventista da Bahia (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 12345
Record Dates: First submitted 2017-05-25; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-04

CONDITIONS: Obesity; Motor Activity; Fatty Acids; Lipid
Keywords: Obesity; Motor Activity; Fatty acids; Lipid
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Will be included 66 women, randomly divided into two groups, control and experiment, overweight, sedentary and aged 18-30 years. After a 12-hour fast, baseline blood collection will be performed in both groups. The experiment group, 12 hours after the first collection, will be submitted to a physical exercise session with energy expenditure of 250Kcal. The volunteers in the control and experiment group will make a second blood collection 24 hours after the first one.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison of fatty acids before and after exercise (Experimental)
  Interventions: Other: Exercise
- Comparison of fatty acids at baseline and 24 hours after (No Intervention)

INTERVENTIONS:
Other: Exercise — After a 12-hour fast, volunteers will collect blood in the antecubital vein to measure basal serum values. 12 after the first blood collection they will perform a physical exercise session on a treadmill. The same will be divided in 3 times: heating, conditioning and cooling. The heating will be of 7 minutes, the cooling of 5 minutes and the time of conditioning will correspond to the energy expenditure of 250Kcal with light intensity based on Borg's perception of effort, that is, in the original scale a value between 9 and 11. After 24 hours after the first blood collection the volunteers will return to the laboratory after a 12-hour fast and blood samples will be collected again.
  Arms: Comparison of fatty acids before and after exercise

SUMMARY:
Introduction: The metabolism of fatty acids in plasma is modulated by their availability in plasma. Individuals with increased weight have increased plasma fatty acids and physical exercise seems to favor the metabolic responses of fatty acid mobilization. Objective: To test the hypothesis that the physical exercise of acute way changes the fatty acids of medium chain of the serum of individuals with increase of the corporal weight. Method: Including 66 women, randomly divided into two groups, control and experiment, overweight, sedentary, and between 18 and 30 years of age. After a 12-hour fast, basal blood collection will be performed. The experiment group, 12 hours after the first collection, will be submitted to a physical exercise session with energy expenditure of 250Kcal. The volunteers in the control and experiment group will make a second blood collection 24 hours after the first one. The fatty acids will be dosed: pelargonic, azelaic, elaidic and oleic by gas chromatography. Intra and intergroup comparisons will be made using the t test for independent and dependent samples, p <0.05.

DETAILED DESCRIPTION:
Randomized clinical trial with accessible population from the School Clinic of the Adventist Faculty of Bahia, Brazil.

All women enrolled in the Clinical School physiotherapy service with a body mass index (BMI) above 24.9kg / m2 will be invited to participate in the study. Sixty-six volunteers who met the inclusion criteria were: age between 18 and 30 years, BMI> 24.9 kg / m2 and sedentarism included randomly. Women who present cardiovascular disease, metabolic disease, history of alcoholism or smoking, use of lipid-lowering drugs, corticoids, diuretics, beta-blockers, contraceptives, hypothyroidism, parenchymal renal diseases or diabetes mellitus will be excluded.

The women will be divided randomly into two groups, experiment and control, both with 33 volunteers.

Group Exercise After a 12-hour fast, the volunteers will be submitted to a blood collection in the antecubital vein to measure basal serum triglycerides, total and fractioned cholesterol, glycemia and insulin. From the values of Glycemia and insulin the values of the Homa-IR and Homa-Beta index were calculated by the equation proposed by Matthews et al.

After 12 days after the first blood collection, the patients will perform a physical exercise session on a treadmill. The same will be divided in 3 times: heating, conditioning and cooling. The heating will be of 7 minutes, the cooling of 5 minutes and the conditioning time will be the one corresponding to the energy expenditure of 250Kcal with light intensity based on the perception of Borg effort, that is, in the original scale a value between 9 and 11. For A better understanding of this scale will be done prior to the day of the exercise accustoming the volunteers to respond adequately when asked about the intensity of the exercise.

After the physical exercise session they will be instructed to return home and maintain their usual diet. After 24 hours after the first blood collection the volunteers will return to the laboratory after a 12-hour fast and will have blood samples collected again. The diet of the two days before the blood test will be evaluated through the 24-hour food recall.

Group control The women in the control group will be submitted to the same data collection protocol of the experimental group, but will not perform exercise 12h after the first collection and will be instructed not to perform physical exercise in the two days prior to blood collection.

ELIGIBILITY:
Inclusion Criteria:

* women
* Body mass index (BMI) over 24.9kg / m2
* 18-30 years
* Sedentary

Exclusion Criteria:

* cardiovascular disease,
* metabolic disease (diabetes, dyslipidemias)
* history of alcoholism or smoking,
* use of lipid-lowering agents,
* use of corticosteroids,
* uses of diuretics,
* use of beta-blockers,
* use of contraceptives,
* use of hypothyroidism,
* use of parenchymal renal diseases

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Levels of fatty acids in individuals with changes in body weight before in the control and experimental group | 30 days
  After blood collection, the initial step for analysis of fatty acids will be the transesterification of the samples through two steps: extraction and hydrolysis / esterification. Similarly, the 99% purity standards of the fatty acids (Pelargonium, azelaic, Oleic and elaidic will also be transesterified. After the transesterification of the standards and samples, they will be analyzed by gas chromatography.

SECONDARY OUTCOMES:
Plasma levels of clinical variables (lipid profile, glycemic profile, oxidative and inflammatory stress) before and after physical activity. | 3 months
  The following data will be analyzed for total lipid profile (total cholesterol, fractions, triglycerides, TG / HDL), inflammatory (Homa-IR, Homa-Beta, Insulin, Glycemia), oxidative stress (glutathione, ON) before And after physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Ana Marice Prof Teixeira Ladeia, Doctor, Study Director — Bahian School of Medicine and Public Health
Locations (1):
- Djeyne Silveira Wagmacker, Cachoeira, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No
The data will not be available in an individual way, only with general data about the population without any form of identification of the subjects

REFERENCES:
- [Background] Holloway GP, Lally J, Nickerson JG, Alkhateeb H, Snook LA, Heigenhauser GJ, Calles-Escandon J, Glatz JF, Luiken JJ, Spriet LL, Bonen A. Fatty acid binding protein facilitates sarcolemmal fatty acid transport but not mitochondrial oxidation in rat and human skeletal muscle. J Physiol. 2007 Jul 1;582(Pt 1):393-405. doi: 10.1113/jphysiol.2007.135301. Epub 2007 May 3. PMID 17478525
- [Result] Jayewardene AF, Mavros Y, Reeves A, Hancock DP, Gwinn T, Rooney KB. Interactions Between Fatty Acid Transport Proteins, Genes That Encode for Them, and Exercise: A Systematic Review. J Cell Physiol. 2016 Aug;231(8):1671-87. doi: 10.1002/jcp.25281. Epub 2016 Feb 2. PMID 26638980
- [Result] Bradley NS, Snook LA, Jain SS, Heigenhauser GJ, Bonen A, Spriet LL. Acute endurance exercise increases plasma membrane fatty acid transport proteins in rat and human skeletal muscle. Am J Physiol Endocrinol Metab. 2012 Jan 15;302(2):E183-9. doi: 10.1152/ajpendo.00254.2011. Epub 2011 Oct 25. PMID 22028411
- [Result] Barres R, Yan J, Egan B, Treebak JT, Rasmussen M, Fritz T, Caidahl K, Krook A, O'Gorman DJ, Zierath JR. Acute exercise remodels promoter methylation in human skeletal muscle. Cell Metab. 2012 Mar 7;15(3):405-11. doi: 10.1016/j.cmet.2012.01.001. PMID 22405075
- [Result] Jabbour G, Iancu HD, Paulin A, Lavoie JM, Lemoine-Morel S, Zouhal H. Effects of Acute Supramaximal Cycle Exercise on Plasma FFA Concentration in Obese Adolescent Boys. PLoS One. 2015 Jun 15;10(6):e0129654. doi: 10.1371/journal.pone.0129654. eCollection 2015. PMID 26076464
- [Result] Jabbour G, Iancu HD, Paulin A. Effects of High-Intensity Training on Anaerobic and Aerobic Contributions to Total Energy Release During Repeated Supramaximal Exercise in Obese Adults. Sports Med Open. 2015;1(1):36. doi: 10.1186/s40798-015-0035-7. Epub 2015 Oct 20. PMID 26512339
- [Result] Plaisance EP, Mestek ML, Mahurin AJ, Taylor JK, Moncada-Jimenez J, Grandjean PW. Postprandial triglyceride responses to aerobic exercise and extended-release niacin. Am J Clin Nutr. 2008 Jul;88(1):30-7. doi: 10.1093/ajcn/88.1.30. PMID 18614721
- [Result] Chen MJ, Fan X, Moe ST. Criterion-related validity of the Borg ratings of perceived exertion scale in healthy individuals: a meta-analysis. J Sports Sci. 2002 Nov;20(11):873-99. doi: 10.1080/026404102320761787. PMID 12430990
- [Result] Santos RD, Gagliardi AC, Xavier HT, Magnoni CD, Cassani R, Lottenberg AM; Sociedade Brasileira de Cardiologia; Arpadi Faludi A, Geloneze B, Scherr C, Kovacs C, Tomazzela C, Carla C, Barrera-Arellano D, Cintra D, Quintao E, Nakandakare ER, Fonseca FA, Pimentel I, Ernesto dos Santos J, Bertolami MC, Rogero M, Izar MC, Nakasato M, Teixeira Damasceno NR, Maranhao R, Cassani RS, Perim R, Ramos S; Sociedade Brasileira de Cardiologia. [First guidelines on fat consumption and cardiovascular health]. Arq Bras Cardiol. 2013 Jan;100(1 Suppl 3):1-40. No abstract available. Portuguese. PMID 23598539
- [Result] Garelnabi M, Litvinov D, Parthasarathy S. Evaluation of a gas chromatography method for azelaic acid determination in selected biological samples. N Am J Med Sci. 2010 Sep;2(9):397-402. doi: 10.4297/najms.2010.2397. PMID 22558586
- [Result] Miyamoto S, Taylor SL, Barupal DK, Taguchi A, Wohlgemuth G, Wikoff WR, Yoneda KY, Gandara DR, Hanash SM, Kim K, Fiehn O. Systemic Metabolomic Changes in Blood Samples of Lung Cancer Patients Identified by Gas Chromatography Time-of-Flight Mass Spectrometry. Metabolites. 2015 Apr 9;5(2):192-210. doi: 10.3390/metabo5020192. PMID 25859693
- [Result] Magkos F, Wright DC, Patterson BW, Mohammed BS, Mittendorfer B. Lipid metabolism response to a single, prolonged bout of endurance exercise in healthy young men. Am J Physiol Endocrinol Metab. 2006 Feb;290(2):E355-62. doi: 10.1152/ajpendo.00259.2005. Epub 2005 Oct 11. PMID 16219668
- [Result] Thackray AE, Barrett LA, Tolfrey K. High-Intensity Running and Energy Restriction Reduce Postprandial Lipemia in Girls. Med Sci Sports Exerc. 2016 Mar;48(3):402-11. doi: 10.1249/MSS.0000000000000788. PMID 26460628
- [Derived] Wagmacker DS, Petto J, Fraga AS, Matias JB, Mota SKA, Rodrigues LEA, Ladeia AM. Metabolic Reponses to a physical exercise session in women with excess body mass: randomized clinical trial. Lipids Health Dis. 2017 Dec 19;16(1):249. doi: 10.1186/s12944-017-0600-9. PMID 29258520